CLINICAL TRIAL: NCT04416581
Title: A Multi-centre, Randomized, Double-Blind, Double-Dummy, Parallel-Group, Phase 4 Efficacy and Safety Study of P-CAB (Tegoprazan 50 mg Once Daily) Compared With PPI (Rabeprazole 20 mg Once Daily) to Reduce Upper Gastrointestinal Events Including Bleeding and Symptomatic Ulcer Disease
Brief Title: Potassium-Competitive Acid Blocker Versus pROton-Pump Inhibitor for GastroproTECTion Strategies In Patients at High Gastro-Intestinal Bleeding Risk Receiving Antithrombotic Therapy
Acronym: PROTECT-HBR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duk-Woo Park, MD (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Associate Professor, Division of Cardiology, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AMCCV2020-05
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndrome; Myocardial Infarction
Keywords: gastroduodenal ulcer; gastrointestinal hemorrhage; peptic ulcer; acute coronary syndrome; coronary artery stent placement; antiplatelet; anticoagulant therapy; PPI; P-CAB; Proton-pump inhibitors; Potassium-Competitive Acid Blockers
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Peptic Ulcer; Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-CAB 50mg group (Experimental): tegoprazan 50 mg + rabeprazole 20mg placebo, once daily.
  Interventions: Drug: P-CAB 50
- PPI group (Active Comparator): rabeprazole 20mg + tegoprazan 50 mg placebo, once daily.
  Interventions: Drug: PPI

INTERVENTIONS:
Drug: PPI — rabeprazole 20mg + tegoprazan 50 mg placebo, once daily.
  Arms: PPI group
Drug: P-CAB 50 — tegoprazan 50 mg + rabeprazole 20mg placebo, once daily.
  Arms: P-CAB 50mg group

SUMMARY:
The primary aim of this study is to evaluate the efficacy and safety of novel P-CAB (tegoprazan 50 mg once daily) as compared with standard PPI (rabeprazole 20 mg once daily) for protection of GI events in patients with known cardiac and vascular disease receiving chronic use of antithrombotic drugs (either antiplatelets, OAC, and its combinations) who are at high GI bleeding risk. The primary hypothesis is that P-CAB (experimental arm) would non-inferior to PPI (standard arm) with respect to the rate of the primary composite end point of GI events at 12 months after randomization.

DETAILED DESCRIPTION:
Before randomization phase, one lead-in subject (N = 300 patients) will be enrolled to perform safety surveillance of standard-dose tegoprazan (50 mg for 6 months) and to ensure the safety of tegoprazan (safety surveillance phase). Data on lead-in subjects will not be included in the data set used for primary analyses.

The safety of tegoprazan will be estimated SIAEs(Special Interest Adverse Events) as follows; Composite Event

1. liver function abnormalities
2. hypergastrinemia, or
3. enteric infection

Definitions

* liver function abnormality: defined as AST or ALT>3× upper limit of normal or two consecutive measurements of total bilirubin >2 x upper limit of normal
* hypergastrinemia
* enteric infection including C.difficile infection

If there are any new tegoprazan-related findings, it will be considered in the estimation.

If there is no safety concern during safety surveillance phase, investigator-driven, randomized, double-blind, double-dummy, active-controlled, clinical trial (N =3,100 patients) will be subsequently performed (randomization phase).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or older with known cardiac and vascular disease who are receiving chronic use of antithrombotic drugs (either antiplatelets, oral anticoagulant (OAC), and its combinations). Specific clinical conditions that may confer a need for long-term antithrombotic therapy may include documented coronary artery disease (stable or unstable angina, acute coronary syndrome, a history of myocardial infarction, or any coronary revascularization), documented cerebrovascular disease (stroke or transient ischemic attack), known peripheral arterial disease or a history of peripheral arterial revascularization, atrial fibrillation, or valvular heart disease requiring interventions (transcatheter aortic valve replacement or transcatheter mitral-valve repair). Concomitant use of a proton pump inhibitor is strongly recommended in patients receiving aspirin monotherapy, DAPT (dual antiplatelet therapy; aspirin plus any P2Y12 inhibitors), DAT (dual antithrombotic therapy; antiplatelet drug plus OAC), TAT (triple antithrombotic therapy; DAPT plus OAC), or OAC monotherapy (warfarin or direct oral anticoagulants) who are at high risk of GI bleeding in order to reduce the risk of gastric bleed or GI events. Based on clinical guidelines, the use of P2Y12 inhibitor monotherapy (i.e. clopidogrel, ticagrelor, or prasugrel) is not considered in trial enrollment.
2. On the basis of clinical guidelines and expert consensus documents, we defined a study population with an increased risk of gastrointestinal bleeding if they had a least 1 or more criteria of the following characteristics. Eligible patients for randomization must meet at least 1 characteristic of these criteria:

   *Definition of patients who are at high risk of gastrointestinal bleeding
   1. Age ≥65 years
   2. Concomitant use of OAC and any antiplatelet therapy (mono or DAPT) (i.e., DAT or TAT)
   3. Long-term use of oral NSAIDs (non-steroidal anti-inflammatory drugs) or steroids or high-dose NSAID therapy even during a relatively short-term period.
   4. History of prior GI bleeding events at any time
   5. History of a previously complicated ulcer
   6. History of peptic ulcer disease or a previously uncomplicated ulcer
   7. Documented Helicobacter pylori infection
3. Patients who voluntarily participated in the written agreement

Exclusion Criteria:

1. Active bleeding at the time of inclusion or a history of hereditary or acquired hemostatic disorder
2. Any clinical contraindication to using of antithrombotic therapies (antiplatelet agents or OAC)
3. Concurrent use of PPI or P-CAB within 4 weeks before randomization
4. Hemodynamically unstable conditions at the time of inclusion: cardiogenic shock at the time of randomization, refractory ventricular arrhythmias, or congestive heart failure (New York Heart Association class IV).
5. Baseline severe anemia (Hgb <8 g/dl at baseline) or transfusion within 4 weeks before randomization
6. Baseline severe thrombocytopenia (platelet count <50,000/mm3)
7. Renal failure dependent on dialysis or severe renal insufficiency (creatinine clearance <15 ml/min)
8. Severe chronic liver disease (defined as variceal haemorrhage, ascites, hepatic encephalopathy, or jaundice)
9. Hypersensitivity or contraindication to PPI, P-CAB, any of the product components, or substituted benzimidazoles
10. Use of clarithromycin and hypersensitivity to macrolide antibiotics for Helicobacter pylori eradication
11. Concomitant use of clarithromycin with terfenadine, cisapride, astemizole, or pimozide for Helicobacter pylori eradication
12. Systemic treatment with strong CYP 3A4 and p-glycoprotein (P-GP) inhibitors (e.g., systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir)
13. Patients who take atazanavir, nelfinavir, or rilpivirine-containing products (see Drug-Drug interaction section)
14. Clinically significant laboratory abnormality at screening (estimated glomerular filtration rate (eGFR) <15 mL/min or elevated liver enzyme [AST, ALT, ALP, total bilirubin] > 3 times upper normal limit [UNL] or any other condition that, in the opinion of the Investigator, precludes participation in the study
15. Any known or suspected malignancy
16. Patients with non-cardiac co-morbidities with a life expectancy of less than 12 months
17. Patients with active treatment for H-pylori infection
18. Women who are pregnant or breastfeeding or female subjects, premenopausal who are not surgically sterile, or, if sexually active not practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and, for those of childbearing potential, who have a positive pregnancy test at screening
19. Participation in another clinical study within 12 months. However, where at least one or more conditions are satisfied, it could be an exception according to an investigator's discretion;

    1. Participated in the observational study expected no effect on the safety and/or effectiveness evaluation of this trial
    2. Screening failed before any interventional factor is involved
    3. Participated in academic trials like strategic or medical device comparison studies conducted under standard therapy provided that there is no additional risk or a specific procedure to a subject and no interference between this trial and other studies

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3320 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The time from randomization to the first occurrence of a composite endpoint of upper GI clinical events, including during the treatment period | 12 months
  This composite outcome included:
  1. Overt upper gastrointestinal bleeding (confirmed by means of upper endoscopy or computed tomography);
  2. Overt upper gastrointestinal bleeding of unknown origin;
  3. Bleeding of presumed occult gastrointestinal origin with a documented decrease in haemoglobin of ≥ 2 g/dL or decrease in hematocrit ≥ 10% from baseline;
  4. Symptomatic gastroduodenal ulcer (confirmed by means of endoscopy or computed tomography) without evidence of gastrointestinal bleeding;
  5. Persistent pain of presumed gastrointestinal origin (duration ≥ 3 days) with underlying multiple erosive disease (5 or more gastroduodenal erosions confirmed by means of endoscopy);
  6. Gastrointestinal obstruction; or
  7. Gastrointestinal perforation.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any of several different events is observed.

SECONDARY OUTCOMES:
The event rate of overt upper gastrointestinal bleeding (confirmed by means of upper endoscopy or computed tomography) | 12 months
The event rate of overt upper GI bleeding of unknown origin | 12 months
The event rate of bleeding of presumed occult GI origin with the documented decrease in Hgb of≥2g/dL or decrease in hematocrit≥10% from baseline | 12 months
The event rate of symptomatic gastroduodenal ulcer(confirmed by means of endoscopy or computed tomography) without evidence of GI bleeding | 12 months
The event rate of the existence of persistent pain of presumed GI origin(duration ≥ 3 days) with underlying multiple erosive diseases (5 or more gastroduodenal erosions confirmed by means of endoscopy) | 12 months
The event rate of gastrointestinal obstruction | 12 months
The event rate of gastrointestinal perforation | 12 months
The time from randomization to discontinuation of study medication attributed to gastrointestinal signs or symptoms | 12 months
The event rate of gastroesophageal reflux disease, as evidenced by symptomatic endoscopically confirmed erosive esophagitis | 12 months
The event rate of composite cardiovascular safety endpoints | 12 months
  composite cardiovascular safety endpoints including:
  1. death from cardiovascular causes;
  2. myocardial infarction; or
  3. stroke
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.
The event rate of death from cardiovascular causes | 12 months
The event rate of myocardial infarction | 12 months
The event rate of stroke | 12 months
The event rate of any coronary or peripheral revascularization | 12 months
The event rate of all-cause mortality | 12 months
The event rate of any possible side effect of proton pump inhibitor (PPI) or Potassium-competitive acid blocker (PCAB) | 12 months

CONTACTS AND LOCATIONS:
Locations (43):
- South Korea (43):
  - Hallym University Sacred Heart Hospital, Anyang
  - Bucheon Sejong Hospital, Bucheon-si
  - Kosin University Gospel Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Sungkyunkwan University Samsung Changwon Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - Chungbuk National University Hospital, Cheonju
  - Gangwon National Univ. Hospital, Chuncheon
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Inje University Ilsan Paik Hospital, Ilsan
  - Jeonbuk National University Hospital, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Chungnam National University Sejong Hospital, Sejong
  - Bundang CHA Hospital, Seongnam
  - Seoul university Bundang hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SNU Boramae Medical Center, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's hospital, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's hospital, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan
  - Yonsei University Yongin Severance Hospital, Yongin-si

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee J, Park HS, Lee J, Choi KD, Kang DY, Ahn JM, Kim W, Lee JY, Lim YH, Kang SH, Kwon SU, Park H, Choi EK, Hong SJ, Kim BK, Jin ES, Jeong JO, Nam CW, Lee WS, Kim SM, Park KH, Her SH, Shin ES, Choi YJ, Yang TH, Kim SH, Suh JW, Park HC, Yoon YH, Yoon MH, Park SJ, Park DW; PROTECT-HBR Trial. Potassium-competitive acid blocker vs proton-pump inhibitor in patients receiving antithrombotic therapy who are at high risk for gastrointestinal bleeding: Rationale and design of the randomized PROTECT- HBR trial. Am Heart J. 2025 Sep;287:50-60. doi: 10.1016/j.ahj.2025.04.001. Epub 2025 Apr 4. PMID 40188976